CLINICAL TRIAL: NCT05045911
Title: A Novel Endoscopic Barbed-clips Suturing for Mucosal Defect Closure After Endoscopic Submucosal Dissection of Colon
Brief Title: An Endoscopic Barbed-clips Suturing for Colorectal ESD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endo-barbed clips suturing
Record Dates: First submitted 2021-08-17; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic Barbed-clips Suturing (Experimental): Patients will be closed the mucosal defect after colorectal ESD using Endoscopic Barbed-clips Suturing.
  Interventions: Procedure: Endoscopic Barbed-clips Suturing

INTERVENTIONS:
Procedure: Endoscopic Barbed-clips Suturing — Endoscopic Barbed-clips Suturing

SUMMARY:
Endoscopic submucosal dissection (ESD) was developed to allow en bloc resection of colorectal neoplasm. Although colorectal ESD has been widely accepted as a minimally invasive treatment option for early colorectal neoplasm, post-ESD bleeding is one of the major adverse events. After ESD procedure, endoscopists close the defects with devices to prevent complications. A novel endoscopic barbed-clips suturing has been developed to simplify endoscopic closure. In this study, the endoscopic barbed-clips will be evaluated when closing defects in the colon after ESD.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) has emerged as a new endoscopic technique that allows en-bloc resection of GI lesions, irrespective of size. The most common complications of the ESD techniques are bleeding and perforation. Several reports have shown that if prophylactic closure of a mucosal defect with clips would reduce the risk of bleeding following endoscopic intervention by ESD. With the advancements in endoscopic therapy, various techniques for prevention of post-ESD complications have been reported. However, there have some limitations including their inability to close large defects and the complexity of the approaches and the need for expensive equipment to complete the procedure. To address these issues, we have devised a novel endoscopic barbed-clips suturing method for mucosal defect closure after endoscopic submucosal dissection of colon. In this study, we assessed the technical feasibility of this novel technique.

ELIGIBILITY:
Inclusion Criteria:

* aged≥20 years with a single clinically or histologically diagnosed colorectal lesions of 20-50mm eligible for which fulfilled criteria for ESD;

Exclusion Criteria:

* Patients with coagulopathy (platelet count < 5 × 10*4, prothrombin time international normalized ratio > 2,
* medical conditions requiring the continuous use of antithrombotic agents
* prior abdominal surgery or radiation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
The technical success rate | 1 day
  Rate of completely closure of the ESD defect

SECONDARY OUTCOMES:
Endoscopic barbed-clips suturing closure time | 1 day
  The time required to close the defect using endoscopic barbed-clips suturing
Rate of patients reported with bleeding/perforation post-ESD procedure | 7 days
  Conduct follow-ups for risk of bleeding and perforation after closure
Clips used post-ESD | 7 days
  Record number of clips needed to close lesion

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No